CLINICAL TRIAL: NCT00337779
Title: A Multinational, Multicenter, Randomized, Parallel-Group, Double-Blind Study to Compare the Efficacy, Tolerability and Safety of Glatiramer Acetate Injection 40 mg/ml to That of Glatiramer Acetate Injection 20 mg/ml Administered Once Daily by Subcutaneous Injection in Subjects With Relapsing Remitting (R-R) Multiple Sclerosis (MS)
Brief Title: Clinical Trial Comparing Treatment of Relapsing-Remitting Multiple Sclerosis (RR-MS) With Two Doses of Glatiramer Acetate (GA).
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GA/9016 (FORTE)
Record Dates: First submitted 2006-06-14; First posted 2006-06-16 (Estimated); Results first posted 2010-05-14 (Estimated); Last update posted 2011-10-10 (Estimated); Status verified 2011-10

CONDITIONS: Relapsing Remitting Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting | interventions — Glatiramer Acetate

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- glatiramer acetate 40 mg (Active Comparator)
  Interventions: Drug: Glatiramer Acetate (GA) 40 mg
- glatiramer acetate 20 mg (Active Comparator)
  Interventions: Drug: glatiramer acetate 20 mg

INTERVENTIONS:
Drug: Glatiramer Acetate (GA) 40 mg — Glatiramer Acetate Injection 40 mg/ml Daily subcutaneous injection for 12 months
  Other Names: Copaxone®
  Arms: glatiramer acetate 40 mg
Drug: glatiramer acetate 20 mg — Glatiramer Acetate Injection 20 mg/ml Daily subcutaneous injection for 12 months
  Other Names: Copaxone®
  Arms: glatiramer acetate 20 mg

SUMMARY:
Teva is developing a 40 mg/ml GA Injection, administered once daily under the skin, for the treatment of R-R MS. The study drug is a higher dose formulation of Copaxone® (20 mg/ml GA), a marketed medication, approved for the treatment of R-R MS. GA is an immunomodulating drug that has anti inflammatory and neuroprotective properties. The study treatment duration is 12 months.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of confirmed and documented MS defined by the Revised McDonald criteria.
2. Subjects must be of the relapsing-remitting (R-R) type.
3. Subject has experienced prior to screening at least one documented relapse in 12 months or at least 2 documented relapses in the 24 months or one documented relapse between 12 - 24 months with at least 1 documented T1-Gd enhancing lesion in the MRI performed 12 months prior screening.
4. Disease duration for at least 6 months.
5. Ambulatory with converted Kurtzke EDSS score of 0 - 5.
6. Relapse free and stable neurological condition at least for 30 days prior screening.
7. Age - 18-55 (inclusive)

Exclusion Criteria:

1. Previous use of Copaxone (glatiramer acetate)
2. Treatment with corticosteroids within 30 days prior screening or between screening and baseline.
3. Chronic corticosteroids treatment - more than 30 consecutive days.
4. Subject with any clinically significant or unstable medical condition.
5. Subjects participating in any other clinical trial (within 12 weeks prior to screening and thereafter).
6. Known history of sensitivity to Gadolinium and inability to successfully undergo MRI scanning.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1155 (Actual)
Dates: Start 2006-08; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chen Duksin, MD, Study Chair — Teva Pharmaceutical Industries, Ltd.; Giancarlo Comi, Prof, Principal Investigator — Istituto Scientifico Fondazione Centro S. Raffaele

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study was conducted according to laws, regulations and administrative provisions related to implementation of Good Clinical Practice as applicable by legislation directives and Standard Operating Procedures. Subjects entered study after being informed and given time to contemplate consent. Enrollment began September 2006 and completed May 2007
Pre-assignment Details: All subjects underwent evaluations including vital signs (blood pressure, pulse, and temperature,) adverse events, concomitant medications and neurological evaluation prior to study entry.
Period: Overall Study
Arm/Group | Glatiramer Acetate 20 mg | Glatiramer Acetate 40 mg
Started | 586 | 569
Completed | 534 | 490
Not Completed | 52 | 79
Not completed — Withdrawal by Subject | 10 | 12
Not completed — Sponsor decision | 1 | 1
Not completed — Physician Decision | 3 | 6
Not completed — Protocol Violation | 1 | 1
Not completed — Lost to Follow-up | 6 | 5
Not completed — Adverse Event | 28 | 51
Not completed — Pregnancy | 3 | 2
Not completed — Death | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Glatiramer Acetate 20 mg | Glatiramer Acetate 40 mg | Total
Number analyzed (Participants) | 586 | 569 | 1155
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 586 | 569 | 1155
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 36.3 (9.0) | 36.3 (9.0) | 36.3 (9.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 421 | 407 | 828
  Male | 165 | 162 | 327
Region of Enrollment [Number; unit: participants]
  Argentina | 14 | 14 | 28
  Belgium | 0 | 1 | 1
  Canada | 15 | 13 | 28
  Czech Republic | 33 | 34 | 67
  Estonia | 11 | 12 | 23
  Finland | 9 | 7 | 16
  France | 10 | 11 | 21
  Germany | 50 | 48 | 98
  Hungary | 27 | 27 | 54
  Israel | 14 | 14 | 28
  Italy | 47 | 43 | 90
  Latvia | 14 | 14 | 28
  Lithuania | 14 | 14 | 28
  Netherlands | 7 | 6 | 13
  Poland | 36 | 35 | 71
  Romania | 29 | 28 | 57
  Russian Federation | 87 | 88 | 175
  Spain | 23 | 22 | 45
  United Kingdom | 11 | 10 | 21
  United States | 135 | 128 | 263

OUTCOME MEASURES:

1. Primary Outcome: The Rate of Confirmed Relapses During the Double-blind Phase (12 Months).
Description: A confirmed relapse is defined as the appearance of one or more new neurological abnormalities or the reappearance of one or more previously observed neurological abnormalities. This change in clinical state must last at least 48 hours and be immediately preceded by an improving neurological state of at least thirty (30) days from onset of previous relapse.
Time Frame: 12 months
Population: ITT
Measure: Mean (Standard Deviation); unit: Number of relapses per patient
Arm/Group | Glatiramer Acetate 20 mg | Glatiramer Acetate 40 mg
Number analyzed (Participants) | 586 | 569
Number of relapses per patient | 0.28 (0.58) | 0.27 (0.54)
Statistical Analysis 1: Comparison: Glatiramer Acetate 20 mg vs Glatiramer Acetate 40 mg; Test type: Superiority or Other; p = 0.4859, Regression, Poisson; Risk Ratio (RR) = 1.0732, 95% CI 2-sided [0.8799 to 1.3090], Standard Error of Mean 0.1013 — 980 subjects randomized into two arms provide approximately 90% power to detect significant difference between groups of 30% or more in rate of confirmed relapses

2. Secondary Outcome: The Number of New T2 Lesions at Month 12 as Compared to the Baseline Scan.
Description: The analysis of this endpoint was based on the outcome of a contrast derived from a baseline-adjusted Negative Binomial Regression including the number of T1 Gd-enhancing lesions at baseline, the volume of T2 lesions at baseline and (pooled) center as covariates.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: T2 Lesions
Arm/Group | Glatiramer Acetate 20 mg | Glatiramer Acetate 40 mg
Number analyzed (Participants) | 586 | 569
T2 Lesions | 2.87 (6.57) | 2.72 (8.36)

3. Secondary Outcome: The Cumulative Number of T1-Gd Enhancing Lesions at Months 3, 6, 9 and 12 (in the Frequent MRI Cohort-described Below).
Description: The Frequent MRI Cohort was a subset of subjects consisting of 234 subjects, for whom MRI scans were performed at months 0 (baseline), 1, 2, 3, 6, 9 and 12. Analysis of the endpoint was based on the outcome of a contrast derived from a baseline-adjusted Negative Binomial Regression with an "offset" variable employing the log of the porportion of the number of available post-baseline scans to adjust for missing MRI scans (if any) and including the number of T1 Gd-enhancing lesions at baseline and (pooled) center as covariates.
Time Frame: 12 months
Population: Frequent MRI cohort
Measure: Log Mean (Standard Deviation); unit: T1 Enhancing Lesions
Arm/Group | Glatiramer Acetate 20 mg | Glatiramer Acetate 40 mg
Number analyzed (Participants) | 121 | 101
T1 Enhancing Lesions | 2.83 (6.58) | 3.49 (8.19)

ADVERSE EVENTS:
Arm/Group | Glatiramer Acetate 20 mg | Glatiramer Acetate 40 mg
Serious Adverse Events (participants affected / at risk) | 25/586 | 24/569
Other Adverse Events (participants affected / at risk) | 499/586 | 490/569
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Glatiramer Acetate 20 mg (N=586) | Glatiramer Acetate 40 mg (N=569)
Coronary Artery Disease (Cardiac disorders) | 0 (0) | 1 (1)
Myocardial Infarction (Cardiac disorders) | 0 (0) | 1 (1)
Palpitations (Cardiac disorders) | 1 (1) | 0 (0)
Supraventricular Tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 2 (2) | 0 (0)
Abdominal Pain (Gastrointestinal disorders) | 1 (1) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Intestinal Obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Swollen Tongue (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Chest Discomfort (General disorders) | 1 (1) | 0 (0)
Chest Pain (General disorders) | 0 (0) | 2 (2)
Chillls (General disorders) | 1 (1) | 1 (1)
Face Oedema (General disorders) | 0 (0) | 1 (1)
Palatal Oedema (General disorders) | 1 (1) | 0 (0)
Swelling Face (General disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 1 (1) | 0 (0)
Cholecystitis Acute (Hepatobiliary disorders) | 1 (1) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Biliary Dyskinesai (Hepatobiliary disorders) | 0 (0) | 1 (1) — Gallbladder Disorder
Anaphylactic Reaction (Immune system disorders) | 1 (1) | 0 (0)
Anaphylactic Shock (Immune system disorders) | 0 (0) | 1 (1)
Hypersensititvity (Immune system disorders) | 0 (0) | 2 (2)
Bronchitis (Infections and infestations) | 0 (0) | 2 (2)
Candidiasis (Infections and infestations) | 1 (1) | 0 (0) — Fungal Infection
Herpes Zoster (Infections and infestations) | 1 (1) | 0 (0)
Device Related Infection (Infections and infestations) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 1 (1)
Pyelonephritis Chronic (Infections and infestations) | 1 (1) | 0 (0)
Complicated Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Crush Injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Multiple Fractures (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Arteriogram Coronary (Investigations) | 0 (0) | 1 (1) — Diagnostic Procedure
Troponin Increased (Investigations) | 0 (0) | 1 (1) — Laboratory Abnormal
Diabetes Mellitus (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Chondropathy (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) — Arthropathy
Back Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscular Weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Breast Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1)
Fibroadenoma of Breast (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) — Breast Neoplasm
Metastases to Lymph Nodes (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Aphasia (Nervous system disorders) | 0 (0) | 1 (1)
Presyncope (Nervous system disorders) | 0 (0) | 1 (1) — Dizziness
Facial Palsy (Nervous system disorders) | 0 (0) | 1 (1)
Tension Headache (Nervous system disorders) | 1 (1) | 0 (0)
Migraine (Nervous system disorders) | 1 (1) | 0 (0)
Multiple Sclerosis Relapse (Nervous system disorders) | 0 (0) | 1 (1)
Radicular Syndrome (Nervous system disorders) | 0 (0) | 1 (1) — Neuropathy Peripheral
Paraesthesia (Nervous system disorders) | 1 (1) | 1 (1)
Loss of Consciousness (Nervous system disorders) | 0 (0) | 1 (1) — Syncope
Panic Attack (Psychiatric disorders) | 1 (1) | 0 (0) — Agitation
Anxiety (Psychiatric disorders) | 0 (0) | 1 (2)
Psychotic Disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Neophrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 4 (4)
Angioedema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Cholecystectomy (Surgical and medical procedures) | 1 (1) | 0 (0)
Coronary Arterial Stent Insertion (Surgical and medical procedures) | 0 (0) | 1 (1)
Laparoscopy (Surgical and medical procedures) | 1 (1) | 0 (0)
Malignant Breast Lump Removal (Surgical and medical procedures) | 1 (1) | 0 (0)
Mastectomy (Surgical and medical procedures) | 1 (1) | 0 (0)
Oophorectomy (Surgical and medical procedures) | 1 (1) | 0 (0)
Spinal Laminectomy (Surgical and medical procedures) | 1 (1) | 0 (0)
Tonsillectomy (Surgical and medical procedures) | 1 (1) | 0 (0)
Varicose Vein Operation (Surgical and medical procedures) | 1 (1) | 0 (0)
Deep Vein Thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Blood Pressure Increased (Vascular disorders) | 0 (0) | 1 (1) — Hypertension
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5.0% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Glatiramer Acetate 20 mg (N=586) | Glatiramer Acetate 40 mg (N=569)
Nausea (Gastrointestinal disorders) | 33 (41) | 33 (45)
Fatigue (General disorders) | 39 (43) | 41 (44) — Asthenia
Chest Discomfort (General disorders) | 32 (43) | 28 (33)
Injection Erythema (General disorders) | 183 (200) | 196 (231)
Injection Site Bruising (General disorders) | 31 (35) | 21 (22)
Injection Site Irritation (General disorders) | 57 (62) | 42 (47) — Injection Site Inflamation
Injection Site Induration (General disorders) | 46 (47) | 54 (62) — Injection Site Mass
Injection Site Mass (General disorders) | 53 (55) | 63 (70)
Injection Site Swelling (General disorders) | 47 (49) | 55 (58) — Injection Site Oedema
Injection Site Pain (General disorders) | 109 (123) | 99 (112)
Injection Site Pruritus (General disorders) | 90 (95) | 93 (99)
Pain in Extremity (General disorders) | 30 (32) | 19 (23)
Upper Respiratory Tract Infection (Infections and infestations) | 49 (65) | 54 (68)
Nasopharyngitis (Infections and infestations) | 78 (102) | 74 (95) — Pharyngitis
Urinary Tract Infection (Infections and infestations) | 43 (50) | 30 (38)
Back Pain (Musculoskeletal and connective tissue disorders) | 28 (34) | 36 (39)
Headache (Nervous system disorders) | 63 (115) | 68 (113)
Depression (Nervous system disorders) | 23 (24) | 36 (36)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 44 (67) | 54 (79)
Flushing (Vascular disorders) | 26 (42) | 36 (49) — Vasodilatation
Dizziness (Nervous system disorders) | 30 (45) | 26 (29)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor has the right 60 days before submission for publication to review/provide comments. If the Sponsor's review shows that potentially patentable subject matter would be disclosed, publication or public disclosure shall be delayed for up to 90 additional days in order for the Sponsor, or Sponsor's designees, to file the necessary patent applications. In multicenter trials, each PI will postpone single center publications until after disclosure or publication of multicenter data.